CLINICAL TRIAL: NCT00481403
Title: Microarray Analysis in Sperm From Fertile and Infertile Males Without Basic Sperm Analysis Abnormalities
Brief Title: Study of Sperm Molecular Factors Implicated in Male Fertility
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Nicolas Garrido, Director of Andrology IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Other Study IDs: VLC-NG-0506-(1003-C-068-JH)
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Male Infertility
Keywords: Sperm, male fertility, microarrays
MeSH Terms: conditions — Infertility, Male | interventions — Microarray Analysis; Gene Expression Profiling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — After sperm washing, sperm pellet was suspended in trizol and immediately frozen by direct immersion in liquid nitrogen and stored in a nitrogen tank until mRNA extraction.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Microarray analysis — Microarray analysis
Behavioral: Microarray — Microarray

SUMMARY:
Sperm analysis following World Health Organization guidelines is unable to explain the molecular causes of male infertility when basic sperm parameters are within a normal range and women do not present gynaecological pathology.

Subsequently, there is a need for accurate diagnostic tools in this sense and microarray technology applied to sperm analysis emerges as a promising field

DETAILED DESCRIPTION:
Sperm analysis based in sperm count and motility has been employed for the diagnosis of male fertility for several decades. It is an easy, inexpensive and useful tool to determine the fertile status of a male but there is still a significant number of infertile males with normal sperm features, as determined by the basic sperm analysis, while they remain unable to reach a full-term pregnancy (1). This fact clearly indicates the need to develop new male infertility tests and accurately diagnose the sperm samples from these individuals.

Recent investigations about sperm mRNA contents have described the relevance of the sperm mRNA stock in fertilization and early embryo development in several species. (2) Although sperm is a quiescent cell from the translational point of view, several functional mRNAs that will be delivered into the oocyte after fertilization, that were synthesized in an earlier phase of the spermatogenesis process can be found (3, 4).

The fertile male transcriptome (stock of mRNAs within the sperm of a male able to have progeny) has been already described (5, 6), confirming the expression of thousands of sequence tags with different intensity of expression.

Moreover, several investigations have demonstrated that a differential expression of some key mRNAs is found in infertile males in comparison with fertile males (1, 7).

Nevertheless, there is no information available neither about the characteristics of the stock sperm mRNAs on infertile males or the differences between fertile and infertile men, although several authors have hypothesized that sperm microarray analysis will be the future in the male infertility diagnosis (2, 8-11).

Microarray technology provides information about a wide range of mRNAs expression within a single experiment, permitting to analyze complete sperm expression profiles (SEP) in cells or tissues. Bioinformatics can help in the organization of such amount of results by following logical processes of gene expression grouping, and analyzing statistically these findings.

Our aim with this work was to compare the SEP in spermatozoa obtained from males with idiopathic infertility versus those from sperm donors of proven fertility by employing microarray technology followed by a functional analysis, in order to determine the genes, sequences and biological processes involved in the sperm physiology that are different in infertile vs. fertile males.

ELIGIBILITY:
Inclusion Criteria:

* Fertile (controls) or infertile males, with sperm parameters above the WHO criteria values

Exclusion Criteria:

* Well established infertility causes

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertile male undergoing assisted reproduction technique without abnormal sperm parameters described by the OMS. Female partners are under 37 years old, IBM lower than 30 kg/m2 and do not present any obvious infertility problem as fallopian tubal obstruction, endometriosis, ovarian failure or polycystic ovarian syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Sperm mRNAs expression profile in samples achieving pregnancy vs those who failed in different assisted reproduction techniques | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Garrido, PhD, Principal Investigator — Instituto Universitario IVI
Locations (1):
- Instituto Universitario Ivi, Valencia, Spain

REFERENCES:
- [Background] 1. Garrido N, Meseguer M, Alvarez J, Simon C, Pellicer A, Remohi J. Relationship among standard semen parameters, glutathione peroxidase/glutathione reductase activity, and mRNA expression and reduced glutathione content in ejaculated spermatozoa from fertile and infertile men. Fertil Steril. 2004 Oct;82 Suppl 3:1059-66. 2. Krawetz SA. Paternal contribution: New insights and future challenges. Nat Rev Genet. 2005;6:633-42. 3. Kramer JA, Krawetz SA. RNA in spermatozoa: Implications for the alternative haploid genome. Mol Hum Reprod. 1997;3:473-8. 4. Wykes SM, Visscher DW, Krawetz SA. Haploid transcripts persist in mature human spermatozoa. Mol Hum Reprod. 1997; 3:15-9.